CLINICAL TRIAL: NCT05293977
Title: Short-Term Use of Antibiotics and Adherence Level: A Randomized Controlled Clinical Trial
Brief Title: Short-Term Use of Antibiotics and Adherence Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: 536/2019
Record Dates: First submitted 2022-01-27; First posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Acute Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Patients in the control group received routine care by the dispensing pharmacist and seen by research assistant for data collection only
  Interventions: Behavioral: Routine care by the dispensing pharmacist
- Intervention (Experimental): Patient in the intervention group was verbally provided with pharmaceutical education/counseling about his/her prescribed antibiotic.
  Interventions: Behavioral: Pharmaceutical education/counseling about prescribed antibiotic

INTERVENTIONS:
Behavioral: Routine care by the dispensing pharmacist — Patients in the control group received routine care by the dispensing pharmacist and seen by research assistant for data collection only
  Arms: Control
Behavioral: Pharmaceutical education/counseling about prescribed antibiotic — Patient in the intervention group was provided with pharmaceutical education about his/her prescribed antibiotic by the trained clinical pharmacist. To prepare the education about antibiotics, the 10 most commonly prescribed antibiotics were determined in advance from hospital records: Amoxicillin or Amoxicillin/Clavulanic acid, Ciprofloxacin, Levofloxacin, Azithromycin, Cefuroxime, Cephalexin, Clindamycin, Doxycycline, Metronidazole, Trimethoprim/Sulfamethoxazole. Standard education points about antibiotics include (i) mechanism of action and/or use, (ii) correct administration method, (iii) correct timing, (iv) possible adverse effect and self-management intervention methods when faced with side effects, (v) what to do in case of missing any dose.
  Arms: Intervention

SUMMARY:
Objectives: To evaluate the impact of educational intervention on antibiotic short-term adherence .

Methods: A prospective randomized controlled study was conducted in a tertiary hospital in Jordan. Adult patients who had an acute infection diagnosis and were prescribed antibiotic pills for short term (< 30 day) at home were included in the study. Patients were recruited and randomly allocated into one of the two groups; control and intervention. Each patient in the intervention group was provided with pharmaceutical education about prescribed antibiotic.

DETAILED DESCRIPTION:
A prospective, single blinded, randomized controlled study was conducted at King Abdullah University Hospital (KAUH) in Jordan. The study was carried out during Aug 2020 till Sep 2021. The primary outcome determined in this study was the impact of pharmaceutical care on the level of short-term adherence among adult patients. An ethical approval was granted from Institutional Review Board in Jordan University of Science and Technology (Ref number 15/126/2019). A sample of 279 patients per each group was required to detect 15% difference in adherence level between intervention and control group at 95% statistical power and at 5% significant level.

All eligible adult patients attending outpatient clinics at KAUH were invited to participate in the study. Adult patients (≥18-year-old) who had an acute infection diagnosis confirmed by a consultant and were prescribed antibiotic pills for short course treatment (< 30 day) at home were included in the study. Those patients who were immunocompromised or used antibiotics for prophylactic indications were excluded. A trained clinical pharmacist (research assistant) interviewed the patients in the waiting area of hospital pharmacy to collect the basic information about the prescribed antibiotics and indications. Written informed consents were obtained from all recruited patients.

Patients were recruited and randomly allocated into one of the two groups (ratio 1:1); ordinary care (control) group and intervention group. Randomization using a simple technique was adopted; even number was assigned for intervention and odd number for control. Each patient in the intervention group was verbally provided with pharmaceutical education/counseling about his/her prescribed antibiotic. The research assistant was responsible for randomization, enrolment and assignment of patients into study groups (intervention Vs control), providing pharmaceutical education about prescribed antibiotics for intervention group and follow up phone calls for both groups. The patients themselves did not know whether they were enrolled in the intervention or control group. To prepare the education about antibiotics, the 10 most commonly prescribed antibiotics were determined in advance from hospital records: Amoxicillin or Amoxicillin/Clavulanic acid, Ciprofloxacin, Levofloxacin, Azithromycin, Cefuroxime, Cephalexin, Clindamycin, Doxycycline, Metronidazole, Trimethoprim/Sulfamethoxazole. Standard education points about antibiotics include (i) mechanism of action and/or use, (ii) correct administration method, (iii) correct timing, (iv) possible adverse effect and self-management intervention methods when faced with side effects, (v) what to do in case of missing any dose. On the other hand, patients in the control group received routine care by the dispensing pharmacist and seen by research assistant for data collection only. The average time interview for patients was 20-25 min in the intervention group Vs approximately 10 min in the control group.

At baseline, socio-demographics and clinical data of all participants were collected such as age, gender, education, employment, family income, and presence of comorbid disease. In addition, questions related to antibiotic use were asked to the patients in both groups such as how many antibiotics were used, symptoms for using antibiotic, and duration/dosing/times interval. Two days after completing the antibiotics course regimens, patients in both groups were followed up by phone to measure adherence by asking them about i) any missing of doses/days of the prescribed antibiotics (subjective method) and ii) number of untaken/remaining pills (objective method). In addition, the patients were asked about whether they use other resources for antibiotics information and the causes of missing duration/doses. In the current study, the participants were labeled as non-adherent if they failed to follow the duration and/ or number of daily doses as prescribed by the physician. These measurements were used based on previous studies.

Data were analyzed using SPSS (version 23). Number (percentage) and median (interquartile range, IQR) were calculated for categorical and continuous data respectively. Univariate analysis was conducted using chi square for categorical variables and Mann Whitney test for continuous data. Factors that were investigated for adherence included: study group, age, gender, marital status, education, employment, income, comorbidity, total number of doses, days antibiotic prescribed, frequency, use the prescribed antibiotic before, and looking at information related to antibiotics. Variables with p value less than 0.25 in univariate analysis were entered in multivariate logistic regression to calculate odds ratio (OR) and 95% confidence interval (95%CI). Intention to treat analysis approach was used in the current study to consider missing data.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18-year-old)
* Patient who had an acute infection diagnosis confirmed by a consultant
* Patients who were prescribed antibiotic pills for short course treatment (< 30 day) at home

Exclusion Criteria:

* Patients who were immunocompromised
* Patients used antibiotics for prophylactic indications

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 589 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Adherence to short-term antibiotic - measured by subjective (questions) and objective (counting remaining pills) methods. | from 1 week to 4 weeks
  Two days after completing the antibiotics course regimens, patients in both groups were followed up by phone to measure adherence by asking them about i) any missing of doses/days of the prescribed antibiotics (subjective method) and ii) number of untaken/remaining pills (objective method).

CONTACTS AND LOCATIONS:
Overall Officials: Basima Almomani, PhD, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan

REFERENCES:
- [Derived] Almomani BA, Hijazi BM, Al-Husein BA, Oqal M, Al-Natour LM. Adherence and utilization of short-term antibiotics: Randomized controlled study. PLoS One. 2023 Sep 5;18(9):e0291050. doi: 10.1371/journal.pone.0291050. eCollection 2023. PMID 37669277